CLINICAL TRIAL: NCT01821781
Title: A Study of Hematopoietic Stem Cell Transplantation (HSCT) in Immune Function Disorders Using a Reduced Intensity Preparatory Regime
Brief Title: Immune Disorder HSCT Protocol
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201301135
Record Dates: First submitted 2013-03-19; First posted 2013-04-01 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Immune Deficiency Disorders; Severe Combined Immunodeficiency; Chronic Granulomatous Disease; X-linked Agammaglobulinemia; Wiskott-Aldrich Syndrome; Hyper-IgM; DiGeorge Syndrome; Chediak-Higashi Syndrome; Common Variable Immune Deficiency; Immune Dysregulatory Disorders; Hemophagocytic Lymphohistiocytosis; IPEX; Autoimmune Lymphoproliferative Syndrome; X-linked Lymphoproliferative Syndrome
Keywords: Immune deficiency; Immune disorders; Immune dysregulatory; Reduced Intensity; Alemtuzumab; Campath
MeSH Terms: conditions — Severe Combined Immunodeficiency; Granulomatous Disease, Chronic; Bruton type agammaglobulinemia; Wiskott-Aldrich Syndrome; Hyper-IgM Immunodeficiency Syndrome; DiGeorge Syndrome; Chediak-Higashi Syndrome; Common Variable Immunodeficiency; Lymphohistiocytosis, Hemophagocytic; Autoimmune Lymphoproliferative Syndrome; Lymphoproliferative Disorders; Immunologic Deficiency Syndromes; Immune System Diseases | interventions — fludarabine; Thiotepa; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preparative (Experimental)
  Interventions: Drug: Transplant preparative regimen of alemtuzumab, fludarabine, thiotepa, and melphalan

INTERVENTIONS:
Drug: Transplant preparative regimen of alemtuzumab, fludarabine, thiotepa, and melphalan — Between days -23 and -15: alemtuzumab test dose, 3mg IV or SQ Day -14: alemtuzumab, 10mg IV or SQ Day -13: alemtuzumab, 15mg IV or SQ Day -12: alemtuzumab, 20mg IV or SQ Days -8 to -4: fludarabine, 30mg/m2 IV Day -4: thiotepa 4mg/kg IV q 12 hours Day -3: melphalan, 140mg/m2 IV Day 0: stem cell infusion Day +7: G-CSF

SUMMARY:
This study hypothesizes that a reduced intensity immunosuppressive preparative regimen will establish engraftment of donor hematopoietic cells with acceptable early and delayed toxicity in patients with immune function disorders. A regimen that maximizes host immune suppression is expected to reduce graft rejection and optimize donor cell engraftment.

ELIGIBILITY:
Inclusion Criteria:

* </= 28 years of age
* Performance status >/= 40
* DLCO >/= 40%
* LVEF >/=40% or LVSF >/=26%
* Serum creatinine < 2x ULN
* Liver enzymes </= 5x ULN
* Negative pregnancy test
* Suitably matched donor (6/6 matched sib UCB, 8/8 matched sib BM or PBSC, 5-6/6 matched unrelated UCB, 7-8/8 matched unrelated BM, double cord)

Exclusion Criteria:

* Known diagnosis of HIV I/II
* Pregnant or breastfeeding
* Uncontrolled invasive fungal or bacterial infections within 1 month prior to starting alemtuzumab
* Uncontrolled viral infection within 1 week prior to starting alemtuzumab

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-03; Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with donor engraftment | 1 year post transplant

SECONDARY OUTCOMES:
Major Transplant Related Toxicities | 1 years post transplant
Time to neutrophil recovery | within 100 days post transplant
Number of patient with acute GVHD | 180 days post transplant
Number of participants with infectious complications | 2 years post transplant
Time to immune reconstitution | 2 years post transplant
Overall survival | 2 years post transplant
Time to platelet recovery | within 100 days post transplant
Number of patients with chronic GVHD | 2 years post transplant
Disease free survival | 2 years post transplant

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Derived] Bhatt ST, Schulz G, Hente M, Slater A, Murray L, Shenoy S, Bednarski JJ. A single-center experience using alemtuzumab, fludarabine, melphalan, and thiotepa as conditioning for transplantation in pediatric patients with chronic granulomatous disease. Pediatr Blood Cancer. 2020 Jan;67(1):e28030. doi: 10.1002/pbc.28030. Epub 2019 Oct 10. PMID 31599480